CLINICAL TRIAL: NCT02982824
Title: Magnesium Supplementation for Children With Drug Resistant Idiopathic Epilepsy: A Pilot Study
Brief Title: Effect of Magnesium Supplementation for Children With Drug Resistant Idiopathic Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics and Head of Pediatric Neurology Unit, Children's, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU M.S 20/2016
Record Dates: First submitted 2016-11-22; First posted 2016-12-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-12

CONDITIONS: Drug Resistant Epilepsy
Keywords: Children; IQ; Idiopathic epilepsy; Magnesium supplementation; Seizure control; Chalfont score
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Magnesium add-on (Experimental): 20 children with drug resistant epilepsy will receive oral magnesium sulfate 6 ml per day which equivalent to 400 mg elemental magnesium (Yuen & Sander, 2012) for 6 months and their regular antiepileptic drugs.
  Interventions: Dietary Supplement: Magnesium
- Antiepileptic drugs only (Placebo Comparator): 20 children with drug resistant epilepsy will receive their regular antiepileptic drugs and placebo for 6 months.
  Interventions: Drug: Placebo - Concentrate
- Healthy controls (No Intervention): To asses serum magnesium level for comparison with the intervention group.

INTERVENTIONS:
Dietary Supplement: Magnesium — Oral magnesium
  Arms: Magnesium add-on
Drug: Placebo - Concentrate — Placebo will be given
  Arms: Antiepileptic drugs only

SUMMARY:
Effect of oral magnesium sulfate (Mg) supplementation will be studied. Children with drug resistant idiopathic epilepsy following up in Pediatric Neurology Clinic, Ain Shams University, will be randomized to either Mg add-on treatment group or anti-epileptic drugs AEDs alone. Serum magnesium, seizure control and Intelligent quotation (IQ) will be done at base line and after 6 months of treatment.

DETAILED DESCRIPTION:
The Aim of this work was to study the effect of Magnesium as add on therapy on clinical seizure control in drug resistant idiopathic epilepsy and IQ.

ELIGIBILITY:
Inclusion Criteria:

* Children with drug resistant idiopathic epilepsy

Exclusion Criteria:

* Structural, Metabolic, Infectious and Unknown etiology epilepsy
* Any neurological disease other than epilepsy
* Any nutritional disorder
* Any other systemic diseases (including Renal disease, Cardiac arrhythmia)
* Drug intake other than antiepileptic drugs (AED)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Seizure control | 6 months
  Change from base line seizure frequency, severity (Chalfont scale) at 6 months.
IQ improvement | 6-months
  Change from base line IQ (Wechsler Intelligence Scale-Revised for Children and Adults)

CONTACTS AND LOCATIONS:
Overall Officials: Sahar MA Hassanein, PhD. MD, Principal Investigator — Pediatrics, Faculty of Medicine, Ain Shams University
Locations (1):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gontijo-Amaral C, Ribeiro MA, Gontijo LS, Condino-Neto A, Ribeiro JD. Oral magnesium supplementation in asthmatic children: a double-blind randomized placebo-controlled trial. Eur J Clin Nutr. 2007 Jan;61(1):54-60. doi: 10.1038/sj.ejcn.1602475. Epub 2006 Jun 21. PMID 16788707
- [Background] Osborn KE, Shytle RD, Frontera AT, Soble JR, Schoenberg MR. Addressing potential role of magnesium dyshomeostasis to improve treatment efficacy for epilepsy: A reexamination of the literature. J Clin Pharmacol. 2016 Mar;56(3):260-5. doi: 10.1002/jcph.626. Epub 2015 Oct 26. PMID 26313363